CLINICAL TRIAL: NCT05590858
Title: Impact of Glycemic Control on Coronary Inflammation Evaluated by Computed Tomography Pericoronary Fat Attenuation Index in Patients With Acute Coronary Syndrome
Brief Title: Glycemic Control on Coronary Inflammation Evaluated by FAI in ACS
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FAI-DM in ACS
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Inflammation Vascular
Keywords: diabetes mellitus; acute coronary syndrome; coronary inflammation; coronary computed tomography angiography; fat attenuation index
MeSH Terms: conditions — Diabetes Mellitus; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-diabetes: patients without diabetes
- well-regulated diabetes: patients with diabetes and HbA1c ≤ 7%
- poorly regulated diabetes: patients with diabetes and HbA1c > 7%

SUMMARY:
This study aimed to clarify the relationship between blood glucose control and the FAI based pericoronary inflammation in low-risk ACS patients with or without diabetes. The results of this study are expected to provide evidence that quantitative assessment of pericoronary FAI helps monitor the local inflammatory activation in diabetic patients with poor glycemic control, therefore, pericoronary FAI evaluation, as a noninvasive imaging biomarker, plays an important role in early detecting coronary atherosclerosis risk in diabetes and allow timely providing appropriate risk reduction strategies in patients at high risk for future cardiovascular events.

DETAILED DESCRIPTION:
Coronary inflammation has been shown to be a cause of the significantly increased risk of cardiovascular disease (CVD) in diabetic patients. This study aimed to investigate the relationship between coronary local inflammation detected by pericoronary fat attenuation index (FAI) and different blood glucose control levels in low-risk acute coronary syndrome (ACS) patients with or without diabetes.A total of 309 patients with low-risk ACS were included in the analysis. Patients were classified into three groups: non-diabetes, well-regulated diabetes and poorly regulated diabetes, depend on the presence or absence of diabetes and the glycemic control evaluated based on a target HbA1c value of 7%. Pericoronary FAI around the proximal of left anterior descending artery (LAD), left circumflex artery (LCX), and right coronary artery (RCA) were evaluated by CCTA, while systemic inflammatory variables and other biochemical indicators were detected by flow cytometry. The results of this study are expected to provide evidence that quantitative assessment of pericoronary FAI helps monitor the local inflammatory activation in diabetic patients with poor glycemic control, therefore, pericoronary FAI evaluation, as a noninvasive imaging biomarker, plays an important role in early detecting coronary atherosclerosis risk in diabetes and allow timely providing appropriate risk reduction strategies in patients at high risk for future cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* patients exhibited chest pain but troponin negative who suspected of low-risk ACS[17];
* patients underwent CCTA examination before elective coronary angiography;
* patients with at least one significant stenosis (≥50%) in major epicardial vessels based on coronary angiography.

Exclusion Criteria:

* patients with missing preprocedural HbA1c values;
* patients with insufficient image quality for FAI analysis,
* patients with previous history of coronary revascularization or myocardial infarction, or chronic kidney disease requiring hemodialysis, or malignant tumor, or immune system disorders, or statin use within 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: low-risk ACS patients who underwent CCTA examination before elective coronary angiography between January 2019 and December 2020 at Renji Hospital
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
pericoronary Fat attenuation index (FAI) | 2021.1.1-2022.10.31
  The pericoronary FAI was defined as the mean CT attenuation of the pericoronary adipose tissue (-190 to -30 HU).
  Peri-stent FAI was measured around the stent segment of all 3 major epicardial coronary vessels.

SECONDARY OUTCOMES:
Level of hsCRP | 2021.1.1-2022.10.31
level of pro-inflammatory cytokines such as IL-2 and IL-6. | 2021.1.1-2022.10.31

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, Doctor, Principal Investigator — RenJi Hospital
Locations (1):
- Cardiology, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun JT, Sheng XC, Feng Q, Yin Y, Li Z, Ding S, Pu J. Pericoronary Fat Attenuation Index Is Associated With Vulnerable Plaque Components and Local Immune-Inflammatory Activation in Patients With Non-ST Elevation Acute Coronary Syndrome. J Am Heart Assoc. 2022 Jan 18;11(2):e022879. doi: 10.1161/JAHA.121.022879. Epub 2022 Jan 13. PMID 35023363
- [Derived] Jiang J, Yin Y, Li Y, Xu B, Zou Z, Ding S, Pu J. Impact of Glycemic Control on Coronary Inflammation Evaluated by Computed Tomography Pericoronary Fat Attenuation Index in Patients with Acute Coronary Syndrome. Rev Cardiovasc Med. 2023 Jul 14;24(7):203. doi: 10.31083/j.rcm2407203. eCollection 2023 Jul. PMID 39077018